CLINICAL TRIAL: NCT00738140
Title: Lifestyle Intervention to Improve Insulin Sensitivity and Markers of Cardiovascular Risk in Prostate Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthew R. Smith, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-081
Record Dates: First submitted 2008-06-23; First posted 2008-08-20 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Prostate Cancer
Keywords: insulin sensitivity; Diabetes Prevention Program; lifestyle intervention
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Intensive lifestyle intervention based on the Diabetes Prevention Program
  Interventions: Behavioral: Diabetes Prevention Program
- B (No Intervention): Will follow the guidelines for healthy living established by the Food Guide Pyramid and the National Cholesterol Education Program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — 12-lesson program which will cover diet, exercise, and behavior modification.
  Arms: A

SUMMARY:
The purpose of this study is to discover if intensive lifestyle changes (such as diet and increased physical activity) improve the body's sensitivity to insulin, and therefore help prevent diabetes and other cardiovascular disease, in men receiving GnRH hormone therapy for prostate cancer.

DETAILED DESCRIPTION:
* In this study, participants will be divided into two groups. One group will undergo intensive lifestyle changes (Lifestyle Intervention Group) designed by the Diabetes Prevention Group, and the other (Control Group) will follow the guidelines for healthy living established by the Food Guide Pyramid and the National Cholesterol Education Program.
* All visits will take place at the General Clinical Research Center at the Massachusetts General Hospital.
* At the initial visit, the following will be performed: Bionutrition evaluation; Oral Glucose Tolerance Test (OGTT); additional blood work and; Dual Energy X-Ray Absorptiometry (DXA) Scan.
* After the initial visit, visits will be scheduled at 3, 6 and 12 months after and the above procedures will be repeated.
* Participants will be randomized into one of the two study groups. Lifestyle Intervention Group: The goal for participants assigned to this group are to achieve and maintain a weight loss of at least 7% of initial body weight through a healthy low calorie, low fat diet and to engage in physical activity of moderate intensity. Control Group: participants in this group will receive standard nutrition and exercise recommendations from the Food Guide Pyramid and the National Cholesterol Education Program Step 1 diet to reduce body weight and increase physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Current Hormone therapy with GnRH agonist of 3 months or longer
* Overweight or obese (body mass index of 25kg/m2 or greater)
* No other conditions that prevent intensive lifestyle intervention

Exclusion Criteria:

* History of diabetes mellitus requiring drug therapy
* Hemoglobin Aic of 7% or greater
* Symptomatic metastatic disease
* Myocardial infarction within 6 months
* Treatment with anabolic agents or metabolic agents known to affect insulin or glucose levels
* Disease progression according to PSA Working Group Criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of intensive lifestyle modification on insulin sensitivity in men receiving GnRH agonist therapy for prostate cancer. | 1 year

SECONDARY OUTCOMES:
To evaluate the effects of intensive lifestyle modification on other markers of cardiovascular disease risk. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smith, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts